CLINICAL TRIAL: NCT03770559
Title: Minimal Invasive Versus Open Radical Antegrade Modular Pancreatosplenectomy for Left-sided Pancreatic Cancer: a Randomized Controlled Trial
Brief Title: The Therapeutic Evaluation(Both Short-term and Long-term Outcome) of Minimal Invasive Radical Antegrade Modular Pancreatosplenectomy for Left-sided Pancreatic Cancer Patients
Acronym: MIRROR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Beijing Municipal Health Commission (Other Government)
Responsible Party: Principal Investigator, Dai Menghua, Professor, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: daimh-RAMPS; No.2020-1-4011 (Other Grant/Funding Number: Beijing Capital Health Research and DEvelopment of Special)
Record Dates: First submitted 2018-11-24; First posted 2018-12-10 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Pancreatic Cancer; Surgery
Keywords: Radical Antegrade Modular Pancreatosplenectomy(RAMPS); Pancreatic Cancer; Minimal Invasive; ERAS; Disease Free Survival
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: The development of study model was divided into 2 parrallel groups( Minimal Invasive RAMPS vs. Open RAMPS) based on the certain surgical procedure underwent
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open-RAMPS (Active Comparator): Patients with pancreatic cancer treated by traditional open surgery
  Interventions: Procedure: Open RAMPS
- MI-RAMPS (Experimental): Patients with pancreatic cancer treated by laparoscopic surgery
  Interventions: Procedure: Minimal Invasive RAMPS

INTERVENTIONS:
Procedure: Minimal Invasive RAMPS — Eligible patients diagnosed as left-side pancreatic cancer in MI-RAMPS group will be treated by minimal invasive RAMPS surgery
  Arms: MI-RAMPS
Procedure: Open RAMPS — Eligible patients diagnosed as left-side pancreatic cancer in Open-RAMPS group will be treated by open invasive RAMPS surgery
  Arms: Open-RAMPS

SUMMARY:
Pancreatic cancer is regarded as "the king of cancer". It is extremely malignant, with a low sensibility to chemotherapy and radiotherapy, and a poor prognosis. Surgical treatment is very important for pancreatic cancer. Radical antegrade modular pancreatosplenectomy (RAMPS) is a standard method for treating pancreatic cancer at the body and tail of pancreas. In the same surgical approach, the investigators are going to compare and discuss the advantages of laparoscopic and open RAMPS in the RCT study.

DETAILED DESCRIPTION:
Open RAMPS is widely used now to treat pancreatic cancer at the body and tail of pancreas. Meanwhile, laparoscopic surgery is proved to have many advantages in other operations. According to primary retrospective study of open and laparoscopic RAMPS, there was no statistically significant difference in the long-term follow-up situations between these two groups, indicating the safety of both this two surgical approaches. The investigators would like to promote a prospective RCT study, to give more evidences of the superiority of laparoscopic RAMPS.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old and older;
2. Pathology diagnosed as pancreatic adenocarcinoma or suspect cancer mass at the pancreatic body or tail;
3. Patients who are eligible and planned to be performed RAMPS procedure;
4. Resectable or borderline resectable tumor by preoperative evaluation.

Exclusion Criteria:

1. Patients with evidence of distant metastasis or advanced arterial invasion so that are not able to continue radical surgery;
2. ASA≥4；
3. Patients who are not willing to be performed open and/or mi-RAMPS;
4. Not pancreatic adenocarcinoma by posteroperative pathology.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Posteroperative length of stay | Until patients were discharged
  The days between the postoperative day-1 to the date when patient was eligible to be discharged.

SECONDARY OUTCOMES:
Overall Survival | more than 1 year
  DFS means the survival duration after surgery.
Operative time | during the surgery
  Durtion of operation
Estimated blood loss | During the surgery
  blood loss volume during the operation
Postoperative pain | Until patients were discharged
  VAS score to measure the degree of postoperative pain
III-IV grade postoperative complication rate | No less than 3 months.
  The ratio between patients with complication(s) and total patients in each groups.
Disease Free Survival | more than 1 year
  DFS means the survival duration after surgery without any evidence of recurrence and metastasis.
R0 resection | up to approximately 2 weeks
  the margin status of resection specimen

CONTACTS AND LOCATIONS:
Overall Officials: Menghua Dai, M.D., Study Chair — PUMCH
Locations (1):
- Department of General Surgery, Peking Union Medical College Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, China, Beijing, China

IPD SHARING:
Plan to Share IPD: No
IPD is not avaiable, but statistical data is avaiable

REFERENCES:
- [Background] Harrison LE, Klimstra DS, Brennan MF. Isolated portal vein involvement in pancreatic adenocarcinoma. A contraindication for resection? Ann Surg. 1996 Sep;224(3):342-7; discussion 347-9. doi: 10.1097/00000658-199609000-00010. PMID 8813262
- [Background] Jimenez RE, Warshaw AL, Rattner DW, Willett CG, McGrath D, Fernandez-del Castillo C. Impact of laparoscopic staging in the treatment of pancreatic cancer. Arch Surg. 2000 Apr;135(4):409-14; discussion 414-5. doi: 10.1001/archsurg.135.4.409. PMID 10768705
- [Background] Mitchem JB, Hamilton N, Gao F, Hawkins WG, Linehan DC, Strasberg SM. Long-term results of resection of adenocarcinoma of the body and tail of the pancreas using radical antegrade modular pancreatosplenectomy procedure. J Am Coll Surg. 2012 Jan;214(1):46-52. doi: 10.1016/j.jamcollsurg.2011.10.008. PMID 22192922
- [Background] Ome Y, Hashida K, Yokota M, Nagahisa Y, Michio O, Kawamoto K. Laparoscopic radical antegrade modular pancreatosplenectomy for left-sided pancreatic cancer using the ligament of Treitz approach. Surg Endosc. 2017 Nov;31(11):4836-4837. doi: 10.1007/s00464-017-5561-6. Epub 2017 Apr 13. PMID 28409377
- [Background] Cao F, Li J, Li A, Li F. Radical antegrade modular pancreatosplenectomy versus standard procedure in the treatment of left-sided pancreatic cancer: A systemic review and meta-analysis. BMC Surg. 2017 Jun 5;17(1):67. doi: 10.1186/s12893-017-0259-1. PMID 28583142
- [Background] Strasberg SM, Linehan DC, Hawkins WG. Radical antegrade modular pancreatosplenectomy procedure for adenocarcinoma of the body and tail of the pancreas: ability to obtain negative tangential margins. J Am Coll Surg. 2007 Feb;204(2):244-9. doi: 10.1016/j.jamcollsurg.2006.11.002. Epub 2007 Jan 4. PMID 17254928
- [Background] Park HJ, You DD, Choi DW, Heo JS, Choi SH. Role of radical antegrade modular pancreatosplenectomy for adenocarcinoma of the body and tail of the pancreas. World J Surg. 2014 Jan;38(1):186-93. doi: 10.1007/s00268-013-2254-8. PMID 24166024
- [Derived] Dai M, Zhang H, Yang Y, Xiu D, Peng B, Sun B, Cao F, Wu Z, Wang L, Yuan C, Chen H, Wang Z, Tian X, Wang H, Liu W, Xu J, Liu Q, Zhao Y. The effect of minimally invasive or open radical antegrade modular pancreatosplenectomy on pancreatic cancer: A multicenter randomized clinical trial protocol. Front Oncol. 2022 Sep 15;12:965508. doi: 10.3389/fonc.2022.965508. eCollection 2022. PMID 36185308